CLINICAL TRIAL: NCT03704597
Title: Cryotherapy as Prophylaxis Against Oral Mucositis After High-dose Melphalan and Autologous Stem Cell Transplantation for Myeloma: a Randomised, Open-label, Phase 3, Non-inferiority Trial Comparing Two and Seven Hours of Cryotherapy.
Brief Title: Cryotherapy Against Oral Mucositis After High-dose Melphalan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Jan-Erik Johansson, Associate Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sahlgrenska
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Myeloma; Mucositis; Cryotherapy Effect
MeSH Terms: conditions — Neoplasms, Plasma Cell; Mucositis | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7-hour cryotherapy (Active Comparator): Standard of care
  Interventions: Other: cryotherapy
- 2-hour cryotherapy (Experimental): Experimental treatment
  Interventions: Other: cryotherapy

INTERVENTIONS:
Other: cryotherapy — Cooling of oral mucosa

SUMMARY:
In this prospective, randomised, controlled, open-label, Phase III, non-inferiority clinical trial trial patients with a diagnosis of myeloma who were undergoing autologous HSCT were randomised 1:1 to receive cryotherapy for 7 hours or 2 hours . Oral mucositis was evaluated prospectively.

DETAILED DESCRIPTION:
We searched MEDLINE and PubMed with the following phrases: "oral mucositis", "oral toxicity", "cryotherapy", "myeloma", "autologous haematopoietic stem cell transplantation", "randomised trial" and "high-dose melphalan".

Oral mucositis, which is a side effect of high-dose chemotherapy, has a major negative impact on the quality of life and survival of patients who undergoing autologous haematopoietic stem cell transplantation (auto-HSCT). For patients with myeloma cryotherapy gives a significant reduction in oral mucositis. The mechanism of action is suggested to be vasoconstriction that is induced by the cooling of the oral mucosa, thereby protecting it from the cytotoxic effects of the chemotherapy. The therapeutic efficacy of cryotherapy in this setting has been confirmed in several trials, it is currently regarded as the standard of care prophylactic regimen for oral mucositis in patients undergoing auto-HSCT for myeloma. However, the long duration of the treatment (7 hours), as reported in the original, placebo-controlled study in 2006, has been associated with significant discomfort for the patients, with negative consequences for compliance.

Uncontrolled trials have previously tested cryotherapy for less than 7 hours in patients with myeloma who receive auto-HSCT. At the time of the planning of the current study in 2014, those results were not yet confirmed in any randomised trial. However last year a randomised trial was published, showing that 2-hour cryotherapy is equally as effective as 6-hour cryotherapy in preventing oral mucositis in patients with myeloma who are treated with high-dose melphalan. The present prospective, randomised study aimed to investigate whether 2 hours of cryotherapy is as effective as 7 hours of cryotherapy in protecting against oral mucositis those patients who are subjected to high-dose melphalan as a conditioning agent for auto-SCT for myeloma.

ELIGIBILITY:
Inclusion Criteria: myeloma, autologous HSCT -

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-03-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Oral mucositis WHO | day 1-14
  Grades 3-4 oral mucositis

REFERENCES:
- [Derived] Johansson JE, Bratel J, Hardling M, Heikki L, Mellqvist UH, Hasseus B. Cryotherapy as prophylaxis against oral mucositis after high-dose melphalan and autologous stem cell transplantation for myeloma: a randomised, open-label, phase 3, non-inferiority trial. Bone Marrow Transplant. 2019 Sep;54(9):1482-1488. doi: 10.1038/s41409-019-0468-6. Epub 2019 Feb 4. PMID 30718802